CLINICAL TRIAL: NCT05618457
Title: Adjustment of Aminoglycoside Dosing Based on Peak Serum Concentration and Bacterial Minimal Inhibitory Concentration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0557-21-HMO
Record Dates: First submitted 2022-10-30; First posted 2022-11-16 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Aminoglycoside Dosing Based on PK/PD Characteristics
Keywords: Aminoglycosides; Minimal Inhibitory Concentration (MIC); Gram negative; PK/PD; Peak concentration (Cmax)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aminoglycoside dose adjustment (Other): Eligible patients will be assessed for attainment of PK/PD target under standard dosing, dose adjustment to attain target will be proposed where appropriate
  Interventions: Drug: Aminoglycoside dose adjustment

INTERVENTIONS:
Drug: Aminoglycoside dose adjustment — Eligible patients may have the aminoglycoside dose adjusted based on pathogen MIC, to attain the PK/PD target of Cam/MIC~10 (8-12)

SUMMARY:
Aminoglycoside (AG) antibiotics have been in clinical use since the 1960s for treating various infections. The main safety concern related to AG use is nephrotoxicity. Based on validated pharmacokinetic-pharmacodynamic (PK-PD) principles shown to predict efficacy, AG dosing has shifted over the past 2 decades from multiple daily dosing to extended-interval dosing, with concomitant reduction in nephrotoxicity. Currently, AG daily dose is calculated according to the patients' adjusted body weight, assuming a common minimal inhibitory concentration (MIC) value.

We hypothesize that once pathogen identity and actual MIC become available, AG daily doses may be further adjusted, using the same PK-PD indices.

In order to investigate this hypothesis, we are conducting a prospective clinical study in which AG doses will be adjusted based on patient- and pathogen-specific factors, while assessing efficacy and safety.

DETAILED DESCRIPTION:
Intervention for all eligible patients:

calculation of Cmax/MIC based on MIC determination and timely peak level determination performed 30 minutes after the first or second AG dose following pathogen identity and MIC availability (as Individual timely monitoring is essential for individual dose adjustment, this will require one additional blood sample to routine clinical practice). If a peak-level monitoring is not available, Cmax will be assessed using commonly used pharmacokinetic prediction tools (equations/calculators.

1. If Cmax/MIC=8-12 - no intervention (aminoglycoside dose unchanged).
2. If Cmax/MIC>12 - decreasing AG dose accordingly, based on clinical calculators, to achieve target Cmax/MIC~10;
3. If Cmax/MIC<8 - increasing AG dose accordingly, based on clinical calculators, to achieve target Cmax/MIC~10; If the calculated dose is larger than acceptable AG dosing, an infectious diseases physician will be consulted for need for alternative therapy.
4. If AG dose has been adjusted, ascertaining PK/PD target attainment (repeat timely peak level determination following dose adjustment).
5. Monitoring clinical and microbiological course and outcomes:

5.1 Clinical efficacy microbiological and clinical cure, in-hospital mortality 5.2 Safety - renal function during therapy, at end of therapy and at discharge or at day 7 after end of therapy, whichever is earlier. Any deterioration in renal function compared with baseline will be categorized according to the RIFLE criteria.

5.3 Aminoglycoside dosing data (proportion end extent of dose adjustments performed)

ELIGIBILITY:
1. Adult patients (≥18yr)
2. Any infection treated with IV gentamycin or amikacin and approved by the consultant infectious diseases specialist, excluding neurosurgical infections, pneumonia, endocarditis or endovascular infections
3. Normal renal function or mild renal impairment (eGFR≥40ml/min)
4. On extended-interval AG and an expected remaining AG course of at least 4 days
5. At least one microbiological specimen with identification of an AG-susceptible pathogen and MIC determination and
6. Signed informed consent form

Exclusion Criteria:

1. Age<18yr
2. Neurosurgical infections, pneumonia, endocarditis or endovascular infections
3. eGFR<40ml/min
4. Empirical aminoglycoside treatment
5. Non Gram-negative pathogen
6. No MIC available for the pathogen
7. Expected remaining treatment duration of less than 4 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy outcome | up to 1 week after end of therapy
  proportion of patients where treatment failure was suspected and attributed to AG dose reduction
Renal outcome | up to 1 week after end of therapy
  Proportion of patients fulfilling RIFLE criteria (any category) baseline
Renal outcome | up to 1 week after end of therapy
  Mean serum creatinine change at end of therapy vs. baseline
Aminoglycoside dosing outcomes: | up to 1 week after end of therapy
  Proportion of patients where AG dose was adjusted based on PK-PD parameters
Aminoglycoside dosing outcomes: | up to 1 week after end of therapy
  Mean change in AG dose following adjustment

CONTACTS AND LOCATIONS:
Overall Officials: Maya Korem, MD, Principal Investigator — Director, Antimicrobial Stewardship Program
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided
YES